CLINICAL TRIAL: NCT04976062
Title: NIRS-IVUS to Improve Assessment of Coronary Artery Disease Severity in Patients Referred for Transcatheter Aortic Valve Implantation; the IMPACTavi Trial
Brief Title: NIRS-IVUS to Improve Assessment of Coronary Artery Disease Severity in Patients Referred for Transcatheter Aortic Valve Implantation
Acronym: IMPACTavi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Infraredx Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: GE IDE No. T00120
Record Dates: First submitted 2021-07-04; First posted 2021-07-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease; Aortic Stenosis, Severe
Keywords: Transcatheter aortic valve implantation; Near-infrared spectroscopy; Intravascular imaging
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Combined near-infrared spectroscopy and intravascular ultrasound imaging (NIRS-IVUS) — The NIRS-IVUS technique is an intravascular imaging technique, combining morphological information derived from intravascular ultrasound (IVUS) and molecular information on plaque composition, namely its respective lipid-core burden, using spectral differences between cholesterol and collagen, detected by near-infrared spectroscopy (NIRS). A combined NIRS-IVUS pullback results in a color-coded map indicating the probability of lipid-rich plaque presence in yellow, co-registered to the corresponding IVUS cross-sections.

SUMMARY:
The aim of the IMPACTavi prospective cohort study is to test feasibility and safety of clinically indicated intravascular coronary imaging with NIRS-IVUS in addition to routine coronary angiography in patients scheduled for TAVI, to improve assessment of CAD severity in this challenging group of patients.

DETAILED DESCRIPTION:
Concomitant coronary artery disease (CAD) is frequent in patients referred for transcatheter aortic valve replacement (TAVI) and there is evidence for a subsequent prognostic impairment. Percutaneous coronary intervention (PCI) is believed to improve prognosis in selected cases, which is why current guidelines recommend PCI to be considered in case of coronary artery diameter stenosis > 70% in proximal segments. Beyond those cases, selection is hampered by inherent shortcoming of the assessment of CAD severity by angiography alone as well as clinical and complex hemodynamic interactions between both pathologies. In patients with CAD alone, the FDA-cleared near-infrared spectroscopy and intravascular imaging (NIRS-IVUS) dual imaging catheter (Indfraredx, Inc., Bedford, USA) has proven the ability to reliably measure lipid plaque burden as well as to identify patients and plaques at increased risk for future adverse cardiovascular events. NIRS-IVUS imaging offers the unique possibility to improve angiographic CAD severity assessment in patients referred for TAVI, avoiding the influence of hemodynamic interactions and pathophysiological overlap between CAD and severe AS.

The IMPACTavi trial is designed as a prospective, non-randomized cohort study to investigate whether NIRS-IVUS-derived lesion characteristics will allow identification of patients likely to suffer adverse clinical events during clinical follow-up after TAVI. Patients with severe aortic stenosis will be qualified for enrollment if routine coronary angiography during diagnostic workup before TAVI shows evidence of coronary artery disease with at least one native vessel without prior stent implantation and at least one lesion requiring NIRS-IVUS imaging for clinical indications, and if at 30mm of total NIRS-IVUS pullback length in sufficient quality for offline analysis have been obtained. Clinical indication, technique and timing of PCI and TAVI will be at the discretion of the interdisciplinary heart-team. The primary and secondary endpoints will be assessed during clinical follow-up out to 24 months. Findings from NIRS-IVUS imaging will be analyzed on a patient- and lesion-level, in order to evaluate correlations of high- vs. low-risk lesion characteristics to the incidence of patient- and lesion-level MACE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and able to give consent
2. Severe aortic stenosis found eligible for transfemoral TAVI by the multi-disciplinary heart team
3. Angiographic evidence of coronary artery disease with absence of coronary stents in at least one native coronary artery
4. At least 30 mm of total NIRS-IVUS pullback length in sufficient quality for offline analysis of at least one native coronary artery with absence of coronary stents, containing at least one lesion requiring NIRS-IVUS imaging for clinical indications
5. Written, informed consent by the patient or her/his legally-authorized representative for participation in the study
6. In women with childbearing potential a negative pregnancy test is mandatory

Exclusion Criteria:

1. Age < 18years
2. Any clinical contraindications to perform NIRS-IVUS
3. ST-elevation myocardial infarction or cardiogenic shock within 48h prior to enrollment
4. Decompensated aortic valve stenosis requiring emergency TAVI
5. History of coronary artery bypass graft (CABG)
6. Severe renal failure with estimated glomerular filtration rate <20 ml/min
7. Malignancies or other comorbid conditions (resulting in a life expectancy <12 months)
8. Inability to fully cooperate with the study protocol
9. Known allergy towards P2Y12 receptor antagonists
10. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic stenosis referred for TAVI with concomitant coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac events as assessed during clinical follow-up and according to current VARC-definitions | 24 months
  Major adverse cardiac events (MACE) is defined as the composite of all-cause mortality, myocardial infarction, unplanned coronary revascularization and hospital readmission due to acute coronary syndrome

SECONDARY OUTCOMES:
Freedom from NIRS-IVUS-emergent complications as assessed by post-NIRS-IVUS control angiography during initial hospital stay, on average 5 days | initial hospital stay
  NIRS-IVUS-emergent complications are defined as coronary impairment following performance of NIRS-IVUS imaging
Incidence of acute kidney injury according to RIFLE/AKIN-criteria assessed during initial hospital stay, on average 5 days | initial hospital stay
Incidence of major vascular complications according to current VARC-defintions, assessed during initial hospital stay, on average 5 days | initial hospital stay
Incidence of major- or life-threatening bleedings according to current VARC-definitions, assessed during initial hospital stay, on average 5 days | initial hospital stay
Incidence of any stroke according to current VARC-definitions, assessed during initial hospital stay, on average 5 days | initial hospital stay
Incidence of all-cause mortality as assessed during clinical follow-up | 24-months
Incidence of myocardial infarction as assessed during clinical follow-up according to current VARC-definitions | 24 months
Incidence of unplanned coronary revascularization as assessed during clinical follow-up | 24 months
Incidence of hospital readmission as assessed during clinical follow-up | 24 months
Incidence of any coronary revascularization as assessed during clinical follow-up | 24 months
Incidence of hospital readmission due to angina pectoris or equivalent as assessed during clinical follow-up | 24 months
NYHA class as defined by the New York Heart Association Functional Classification assessed at 24-months clinical follow-up | 24 months
CCS class as defined by the Canadian Cardiovascular Society grading of angina pectoris assessed at 24-months clinical follow-up | 24 months
Delta left-ventricular ejection fraction at 3- and 12-months follow-up compared to baseline | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joner, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (2):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided